CLINICAL TRIAL: NCT01329718
Title: Specimen Collection Protocol for the Performance Evaluation of the Septin 9 Assay
Brief Title: Specimens for Septin 9 Performance
Acronym: SPR0012
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Epigenomics, Inc (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Epigenomics_SPR0012
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Colorectal Cancer
Keywords: Stability of the Septin 9 biomarker; Epi Pro Colon Test; CRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- CRC Group (Experimental)
  Interventions: Other: Blood Sample

INTERVENTIONS:
Other: Blood Sample — Blood sample collection

SUMMARY:
Epigenomics has identified methylated gene regions that are specific for colorectal cancer (CRC). Through Epigenomics' marker discovery and validation process Septin 9 was identified as a particularly robust methylation marker for detection of CRC. Epigenomics is currently developing a blood based CRC screening test based on Septin 9 and is performing a large prospective clinical trial showing its clinical utility in a population at average risk for CRC. Parallel to this trial further activities are needed to evaluate, optimize, and develop pre-analytical and analytical workflows as well as molecular assays making possible the use of Septin 9 methylation in the clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older at the time of the blood draw
* Histologically confirmed or strong clinical suspicion of adenocarcinoma of the colon or rectum
* CRC defined as invasive adenocarcinoma

Exclusion Criteria:

* Previous personal history of colorectal cancer
* Any cancer specific treatment (e.g. polypectomy, chemotherapy, radiation, or surgery) prior to blood draw, including neoadjuvant treatment
* Known infection with HIV, HBV or HCV
* Subject concurrently receiving intravenous fluid at the time of the specimen collection

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 562 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the Epi proColon test | 12 months
  The primary objective of the investigation is to determine the safety and effectiveness of the Epi proColon test in precision and reproducibility studies and varying conditions including interfering substances and co-morbidities associated with the testing population. The specimens collected as described in this protocol will be used in the experiments needed to achieve this objective. Validate the Stability of the Septin 9 Biomarker.